CLINICAL TRIAL: NCT03846232
Title: T1rho: Detection of Cerebral Proteinopathy in Alzheimer's Disease Through Magnetic Resonance Imaging
Brief Title: Detection of Cerebral Proteinopathy in Alzheimer's Disease Through Magnetic Resonance Imaging
Acronym: T1rho
Status: Completed | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: T1rho/BBRC2017
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitive impairment. Alzheimer's disease: Diagnosed with AD as defined per the International Working Group IWG 2 criteria (fulfilling core clinical criteria plus positive core AD CSF biomarkers)
  Interventions: Other: No intervention
- Cognitively unimpaired, preclinical Alzheimer's disease: Normal cognition as defined by the ALFA study cognitive workup Positive amyloid PET in the last 30 months
  Interventions: Other: No intervention
- Cognitively unimpaired, control: Normal cognition as defined by the ALFA study cognitive workup Negative amyloid PET in the last 30 months
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The main goal of the T1rho/BBRC2017 study is to assess the capability of the MRI sequences T1rho + multicomponent T2 relaxation analysis of detecting abnormal cerebral protein deposition in AD patients in comparison with an age-matched cognitively healthy control group. Both the AD and control groups will had previously undergone amyloid PET imaging to confirm/discard cerebral proteinopathy in the context of other research studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Informed, written consent form
* To fully satisfy the criteria for one of the two following 2 groups:

  1. for the AD group:

     * Diagnosed with AD as defined per the International Working Group IWG 2 criteria (fulfilling core clinical criteria plus positive core AD CSF biomarkers): Light to mild AD defined by Mini-Mental State Examination (MMSE) score between 15 and 27 (included).
     * Documented positive visual read (as per EMA-approved procedures for each respective tracer) of an amyloid PET scan, which in the opinion of the principal investigator is consistent with a diagnosis of AD in the last 24 months.
     * Lumbar puncture with core AD CSF biomarkers available in the last 24 months.
  2. For the cognitively health group:

     * Normal cognition as defined by the ALFA study cognitive workup (Molinuevo et al. 2016).

CONFIDENTIAL 17

* [18F]-Flutemetamol PET scan performed in the context of the PET FLUTEMETAMOL-FDG/BBRC2015 study in the last 24 months.
* Lumbar puncture with core AD CSF biomarkers preferably available in the last 24 months.

Exclusion Criteria:

* Past or present history of major brain disorders other than MCI or AD.
* Contraindication to MRI scanning or conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
* Participation in a clinical trial for a disease modifying drug for AD.
* Hypoperfusion pattern not consistent with AD diagnosis, as assessed by ASL.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participating subjects are (1) patients with AD with typical presentation for which an amyloid PET is already available or (2) age-matched cognitively healthy adults that, similarly, have available amyloid PET imaging information.
  Specifically, a subsample of 40 cognitively healthy adult participants from the ALFA study [25] (http://clinicaltrials.gov/ct2/show/NCT01835717; Estudi 45-65 FPM/2012) will be selected to undergo the present study on the basis of their cerebral amyloidosis as assessed by PET in the context of the PET FLUTEMETAMOL-FDG/BBRC2015 study (20 negative and 20 positive). AD patients (n=20) will be recruited from collaborating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of abnormal cerebral protein levels | at inclusion
  Discriminant capacity to detect abnormal cerebral protein levels in 3 age-matched groups: cognitively normal subjects without (CN) and with abnormal biomarker levels (PreAD), and Alzheimer Disease patients (AD).

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelonabeta Brain Research Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No